CLINICAL TRIAL: NCT07085754
Title: Effects of Acute Sleep Deprivation on Individuals With Different APOE Genotypes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yuhui Qiu (Other)
Responsible Party: Sponsor-Investigator, Yuhui Qiu, Principal Investigator, Guangdong Provincial Hospital of Traditional Chinese Medicine
Organization: Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: ZF2025-206-01
Record Dates: First submitted 2025-07-06; First posted 2025-07-25 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-07

CONDITIONS: Sleep; Sleep Deprivation
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sleep Deprivation (Experimental): 24 hours of sleep deprivation
  Interventions: Behavioral: Sleep Deprivation
- Control (No Intervention): 24 hours of a normal work-rest schedule

INTERVENTIONS:
Behavioral: Sleep Deprivation — Sleep deprivation for up to 24 hours with no naps or other sleep periods
  Arms: Sleep Deprivation

SUMMARY:
This study aims to investigate the effects of 24-hour acute sleep deprivation on plasma Alzheimer's disease biomarkers and multi-omics in individuals with different APOE genotypes, to elucidate the potential role of acute sleep deprivation in AD risk.

DETAILED DESCRIPTION:
This is a randomized controlled trial designed to enroll 60 healthy volunteers. Stratified randomization will be used, with three strata defined by APOE genotype (APOE ε3/3, APOE ε4 carriers, and APOE ε2 carriers) in a 1:1:1 ratio. Within each stratum, participants will be randomly assigned in a 1:1 ratio to either the acute sleep-deprivation group or the non-acute sleep-deprivation group. The intervention will consist of 24 hours of acute sleep deprivation. The primary outcome measure is the change from baseline in plasma Aβ42 on the first day after randomization.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years, gender not limited
* Healthy (with no clinically significant abnormal findings in the physical examination report or self-reporting as healthy) and not on medications
* Cognitively normal (Mini-Mental State Examination (MMSE) score > 28)
* Sleep duration of 7-9 hours per night, good sleep quality (Pittsburgh Sleep Quality Index (PSQI) ≤ 5 points)
* Written informed consent, voluntarily participate in this study, and be able to cooperate with the physician to complete the clinical study

Exclusion Criteria:

* Presence of day-night sleep reversal
* Shift work within the past 6 months
* Travel across time zones or experience of jet lag within the past three weeks
* Current smoking or nicotine use; alcohol consumption exceeding five standard units per week (one standard alcohol unit is defined as 10 mL [or 8 g] of pure alcohol)
* Consumption of strong tea, coffee, or caffeine-containing foods and beverages within one week before study participation
* Family history of early-onset dementia
* Self-Rating Depression Scale (SDS) score ≥ 53, Self-Rating Anxiety Scale (SAS) score ≥ 50
* Female participants who are currently pregnant or breastfeeding
* Individuals who need to drive or operate vehicles or machinery during the study period

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-08 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Plasma Aβ42 levels | 1 day after randomization

SECONDARY OUTCOMES:
Plasma Aβ40 levels | 1 day after randomization
Plasma t-tau levels | 1 day after randomization
Plasma p-tau181 levels | 1 day after randomization
Plasma p-tau217 levels | 1 day after randomization
Plasma NfL levels | 1 day after randomization
Plasma GFAP levels | 1 day after randomization
Plasma Aβ42/Aβ40 levels | 1 day after randomization
Plasma t-tau/Aβ42 levels | 1 day after randomization
Plasma p-tau181/Aβ42 levels | 1 day after randomization
Plasma p-tau217/Aβ42 levels | 1 day after randomization
Fatigue Scale-14 | 1 day after randomization
  The Fatigue Scale-14 has a minimum score of 0 and a maximum score of 33; higher scores indicate greater fatigue severity.
Positive and Negative Affect Schedule | 1 day after randomization
  The Positive and Negative Affect Schedule comprises two subscales: Positive Affect and Negative Affect. Each subscale ranges from 10 to 50, with higher scores indicating greater accumulation of the corresponding affect.
N-back tasks | 1 day after randomization
  N-back test, participants are required to identify target digits that match the stimuli presented N steps earlier on the screen

OTHER OUTCOMES:
PET/MRI | 1 day after randomization
  Assessed using Positron Emission Tomography/Magnetic Resonance Imaging(PET/MRI)
Proteomics | 1 day after randomization
  The plasma proteomics will be determined by Liquid Chromatography - MassSpectrometry
Metabolomics | 1 day after randomization
  The plasma metabolomics will be determined by Liquid Chromatography - MassSpectrometry

CONTACTS AND LOCATIONS:
Locations (1):
- Guangdong Provincial Hospital of Chinese Medicine, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No